CLINICAL TRIAL: NCT02347865
Title: Prospective Observational Study to Describe Characteristics and Management of Postmenopausal Women With Osteoporosis Treated With Prolia® in France and Its Use in Routine Clinical Practice
Brief Title: Characteristics and Management of Postmenopausal Women With Osteoporosis Treated With Prolia® in France
Acronym: PILOTE
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20130240
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Post Menopausal Osteoporosis
Keywords: osteoporosis post menopausal women
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- wave 1: postmenopausal women with osteoporosis treated with Prolia
  Interventions: Drug: AMG 162 - Prolia
- wave 2: postmenopausal women with osteoporosis treated with Prolia
  Interventions: Drug: AMG 162 - Prolia

INTERVENTIONS:
Drug: AMG 162 - Prolia — 500 patients
  Other Names: denosumab
  Groups: wave 1
Drug: AMG 162 - Prolia — 250 patients, one year later
  Other Names: denosumab
  Groups: wave 2

SUMMARY:
The purpose of the study is to describe the characteristics and management of post menopausal women with osteoporosis treated with Prolia in France, and examine the use of Prolia in routine clinical practice in France

DETAILED DESCRIPTION:
This is a multicenter, observational and non-interventional study in PMO patients who receive Prolia® (60 mg subcutaneous [SC]) in France. Patients in the study will be enrolled in 2 waves, each targeting specific aspects of the overall study objectives. The first wave will enroll approximately 500 patients who will be followed for approximately 30 months from the first injection. Patients enrolled in this wave will provide descriptive data on persistence to Prolia® as well as a description of the characteristics of patients being prescribed Prolia®, information regarding Prolia® prescription and administration, procedures pertaining to Prolia® and safety.

The second wave will enroll approximately 250 patients and will only provide a cross-sectional description of the characteristics of patients being prescribed Prolia.

Around 2000 specialists in rheumatology and 9000 general practitioners will be randomly selected from a list of rheumatologists whether in hospital or private practice nationwide and a list of general practitioners managing patients with osteoporosis.

In all, 300 physicians initially interested to participate are expected, from which about 180 physicians will be qualified to participate. One-hundred and ten physicians will be initiated.

There are no procedures or changes to the routine clinical management of patients participating in the study. Baseline characteristics will be described for patients enrolling in both waves 1 and 2. Patients enrolling in wave 1 will be followed for approximately 30 months from the date of first injection in the study. It is anticipated that patients will return to the site. Clinical information obtained for routine clinical practice will be recorded where available, including Prolia administration, previous and current therapies, medical history (including fracture), ADRs, SADRs and co-morbidities.The study is descriptive in nature, and no formal hypothesis will be tested. In general, data summaries will be presented by wave and by subgroups of interest.

ELIGIBILITY:
Inclusion Criteria:

* post menopausal osteoporosis women in whom a decision has been made to treat with Prolia in the last 4 weeks
* received their first prescription of Prolia in the last 4 weeks
* patient has provided informed consent before enrolling in the study

Exclusion Criteria:

* patients participating in ongoing or previous Denosumab clinical trials

Ages: 40 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post menopausal women with osteoporosis, treated with Prolia
Sampling Method: Probability Sample
Enrollment: 777 (Actual)
Dates: Start 2015-06-16 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
patient occurence of persistence (persistence is defined in the outcome description) at 12 months | 12 months
  To evaluate the persistence with Prolia at 12 months in post menopausal women with osteoporosis (PMO) in France. To evaluate the persistence with Prolia at 24 months in PMO women in France. Patients will be defined as persistent with Prolia at 12 months if the patient receives at least 2 injections and the second injection at 6 months is no later than 6 months + 8 weeks (or 239 days) from the baseline injection

SECONDARY OUTCOMES:
patient occurence of persistence (persistence is defined in the outcome description) at 24 months and time to non-persistence at 24 months | 24 months
  To evaluate the persistence with Prolia at 24 months in PMO women in France. Patients will be defined as persistent with Prolia at 24 months if the patient receives at least 4 injections (including the baseline) and the time between any 2 injections is not more than 6 months + 8 weeks (or 239 days)
describe the use of Prolia in routine clinical practice during approximately 30 months from the first injection | 30 months from first injection
  to describe the occurence of patients referred to another physician for follow up on prolia treatment, the number of injections received by the patient, the occurence of a patient receiving the first, second, third, fourth and fifth injections, the number of times a patient received Prolia injection by the prescriber and the number of times a patient received a Prolia injection outside the prescriber's office by nurse or other healthcare provider
patient occurence of Adverse Drug Reactions (ADRs) and Serious Adverse Drug Reactions (SADRs) as collected in routine clinical practice | 30 months or early termination
  to describe the patient occurence of ADRs and SADRs as collected in routine clinical practice
Occurrence of patient reported osteoporosis related vertebral and non vertebral fractures reported during the study | 30 months or early termination
  Patient occurence of osteoporosis related vertebral and non vertebral fractures during the study. Osteoporosis related fractures are defined as all fractures excluding skull, facial bones, mandible, metacarpus, finger phalanges, toe phalanges and cervical vertebrae and not associated with known high trauma severity or pathological fractures.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Amgen, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com